CLINICAL TRIAL: NCT04556201
Title: A Prospective, Multicenter, Post-Market Clinical Registry to Collect Real-World Evidence on the Clinical Performance of the SOLTIVE™ Laser for Treatment of Kidney or Ureteral Stones
Brief Title: The Performance of the SOLTIVE Laser System for Laser Lithotripsy in Kidney or Ureteral Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-URO-01
Record Dates: First submitted 2020-09-07; First posted 2020-09-21 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Kidney Stone; Ureteral Stone
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Thulium Fiber Laser lithotripsy (Experimental): Subjects who have a medical indication for ureteroscopy, percutaneous nephrolithotomy (PCNL) or mini PCNL
  Interventions: Device: SOLTIVE™ Premium SuperPulsed Laser Fiber System

INTERVENTIONS:
Device: SOLTIVE™ Premium SuperPulsed Laser Fiber System — SOLTIVE™ SuperPulsed Laser Fiber System and SOLTIVE™ Laser Fibers for single-use only

SUMMARY:
The purpose of this study is to collect real-world evidence on the performance of the SOLTIVE™ Premium SuperPulsed Laser System for laser lithotripsy in ureteroscopy, percutaneous nephrolithotomy (PCNL) and mini PCNL for kidney and ureteral stones.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Medical indication for ureteroscopy, percutaneous nephrolithotomy (PCNL) or mini PCNL
3. Willing and able to provide informed consent
4. Female and of childbearing age with a negative pregnancy test

Exclusion Criteria:

1. Contraindicated for uteroscopy, PCNL or mini PCNL as determined by the physician
2. Inability to tolerate anesthesia for any reason
3. Unable or unwilling to provide informed consent
4. Concurrently participating in another competing clinical study
5. Known ureteral stricture
6. Unwilling or unable to return for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Stone free rate | 3 month
  Stone free rate as determined by standard of care imaging

SECONDARY OUTCOMES:
Total laser energy time | During procedure
  Measured from first to last footswitch press in minutes
Total procedure time | During procedure
  Measured from time of initial ureteroscope insertion to time of ureteroscope withdrawal in minutes
Accessory devices used | During procedure
  Types of accessory devices used during the procedure (ureteroscopy, PCNL or mini-PCNL) and the total time used during the procedure in minutes
Adverse events | At procedure, immediate post-procedure, 1 month follow-up and 3 month follow-up
  AEs related to device or procedure and non-serious AEs related to device or procedure
Device deficiencies | During procedure
  Number of device deficiencies during the procedure
Rate of treatment/interventions needed | At 1 month follow-up and 3 month follow-up
  Types of treatments and/or interventions needed post-procedure at the follow-up visits and the number of times treatments and/or interventions were performed

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — University of British Columbia; Olivier Traxer, MD, Principal Investigator — Tenon Hospital, Sorbonne University, Paris
Locations (7):
- United States (5):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Kansas University Medical Center, Kansas City, Kansas
  - Mount Sinai West, New York, New York
  - Ohio State Wexner Medical Center, Columbus, Ohio
- University Southern Denmark, Fredericia, Denmark
- Hospital CUF Descobertas, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Subject data collected during the study after de-identification.
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication

REFERENCES:
- [Result] Sorokin I, Mamoulakis C, Miyazawa K, Rodgers A, Talati J, Lotan Y. Epidemiology of stone disease across the world. World J Urol. 2017 Sep;35(9):1301-1320. doi: 10.1007/s00345-017-2008-6. Epub 2017 Feb 17. PMID 28213860
- [Result] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Result] C. Türk, A. Skolarikos, A. Neisius, A. Petrik, C. Seitz, K. Thomas, EAU Guidelines. European Association of Urology (EAU). 2019.
- [Result] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART I. J Urol. 2016 Oct;196(4):1153-60. doi: 10.1016/j.juro.2016.05.090. Epub 2016 May 27. PMID 27238616
- [Result] Aldoukhi AH, Knudsen BE, Black KM, Hall TL, Roberts WW, Ghani KR. Are We Cutting Ourselves Short? Laser Lithotripsy Performance Based on Differences in Fiber-tip Preparation. Urology. 2019 Dec;134:79-83. doi: 10.1016/j.urology.2019.08.027. Epub 2019 Aug 30. PMID 31476349
- [Result] Peter Kronenberg, Olivier Traxer. V1718 laser fibers, pulse energy and retropulsion- what we can see and what we can´t. ResearchGate. 2013.
- [Result] Humphreys MR, Shah OD, Monga M, Chang YH, Krambeck AE, Sur RL, Miller NL, Knudsen BE, Eisner BH, Matlaga BR, Chew BH. Dusting versus Basketing during Ureteroscopy-Which Technique is More Efficacious? A Prospective Multicenter Trial from the EDGE Research Consortium. J Urol. 2018 May;199(5):1272-1276. doi: 10.1016/j.juro.2017.11.126. Epub 2017 Dec 16. PMID 29253579
- [Result] Sofer M, Watterson JD, Wollin TA, Nott L, Razvi H, Denstedt JD. Holmium:YAG laser lithotripsy for upper urinary tract calculi in 598 patients. J Urol. 2002 Jan;167(1):31-4. doi: 10.1016/s0022-5347(05)65376-1. PMID 11743269
- [Result] Zarrabi A, Gross AJ. The evolution of lasers in urology. Ther Adv Urol. 2011 Apr;3(2):81-9. doi: 10.1177/1756287211400494. PMID 21869908
- [Result] Kronenberg P, Somani B. Advances in Lasers for the Treatment of Stones-a Systematic Review. Curr Urol Rep. 2018 May 17;19(6):45. doi: 10.1007/s11934-018-0807-y. PMID 29774438
- [Result] Traxer O, Keller EX. Thulium fiber laser: the new player for kidney stone treatment? A comparison with Holmium:YAG laser. World J Urol. 2020 Aug;38(8):1883-1894. doi: 10.1007/s00345-019-02654-5. Epub 2019 Feb 6. PMID 30729311
- [Result] Scott, N. J., C. M. Cilip, and N. M. Fried. Thulium Fiber Laser Ablation of Urinary Stones Through Small-Core Optical Fibers, IEEE Journal of Selected Topics in Quantum Electronics. 2009;(15):435-40.
- [Result] Pasqui F, Dubosq F, Tchala K, Tligui M, Gattegno B, Thibault P, Traxer O. Impact on active scope deflection and irrigation flow of all endoscopic working tools during flexible ureteroscopy. Eur Urol. 2004 Jan;45(1):58-64. doi: 10.1016/j.eururo.2003.08.013. PMID 14667517
- [Result] Kronenberg P, Traxer O. The truth about laser fiber diameters. Urology. 2014 Dec;84(6):1301-7. doi: 10.1016/j.urology.2014.08.017. PMID 25432821
- [Result] Mahmood SN, Toffeq H, Fakhralddin S. Sheathless and fluoroscopy-free retrograde intrarenal surgery: An attractive way of renal stone management in high-volume stone centers. Asian J Urol. 2020 Jul;7(3):309-317. doi: 10.1016/j.ajur.2019.07.003. Epub 2019 Jul 16. PMID 32742931
- [Result] Enikeev D, Taratkin M, Klimov R, Alyaev Y, Rapoport L, Gazimiev M, Korolev D, Ali S, Akopyan G, Tsarichenko D, Markovina I, Ventimiglia E, Goryacheva E, Okhunov Z, Jefferson FA, Glybochko P, Traxer O. Thulium-fiber laser for lithotripsy: first clinical experience in percutaneous nephrolithotomy. World J Urol. 2020 Dec;38(12):3069-3074. doi: 10.1007/s00345-020-03134-x. Epub 2020 Feb 27. PMID 32108256